CLINICAL TRIAL: NCT04464720
Title: AIM to Improve Asthma: Airflow Improvements During Meal-Prep
Acronym: AIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-01-10615; R21ES030173 (NIH)
Record Dates: First submitted 2019-12-18; First posted 2020-07-09 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-09

CONDITIONS: Asthma in Children; Pollution; Exposure
Keywords: asthma; pediatric; indoor air pollution; particulate matter; nitrogen dioxide; cooking; ventilation
MeSH Terms: conditions — Asthma; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: This is a trial with a single group, where they receive the intervention following one week of baseline data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention after One Week (Other): This arm will have baseline data on air pollutant levels, stove use and range hood use collected for one week prior to receiving an educational intervention aimed at increasing use of the range hood. Data following the intervention will be collected for an additional week.
  Interventions: Behavioral: Cooking Ventilation Intervention

INTERVENTIONS:
Behavioral: Cooking Ventilation Intervention — An educational video presentation for the families regarding the importance of ventilation use during and after cooking, and strategies for improving the ventilation during cooking, has been created by Dr. Holm, with input from Youth Research Assistants (YRAs) The youth involvement will help to ensure that the information is presented in a way that will resonate with the local community and will also provide the youth with exposure to developing health education tools. The educational video will be shown to families at the time of the intervention visit and they will receive printed reminder materials of what they have learned.

SUMMARY:
The investigators propose a pilot trial of kitchen ventilation in the homes of children using a youth engaged research strategy.

DETAILED DESCRIPTION:
In this trial of children ages 6-12, children and their households will receive an intensive home kitchen ventilation intervention after one week of baseline data collection. The intervention includes education regarding improving ventilation in their homes during cooking and replacement of their range hood if it has inadequate flow or an intolerable noise level. During baseline data collection periods the households will be encouraged to continue their regular cooking patterns. The investigators will measure home particulate matter <2.5 microns (PM2.5) and nitrogen dioxide (NO2) levels for one week at baseline, and a final week after all remaining families receive the cooking ventilation intervention, to assess for changes within each household. The investigators will also examine changes in airways inflammation (as measured by the exhaled fraction of nitric oxide, FeNO), lung function (as measured by spirometry), and reported symptoms after the baseline and intervention period. Members of the research team have successfully conducted youth participatory action research in the low-income, high asthma prevalence community of Richmond, California (CA) as well as extensive youth participatory action research on other environmental health concerns in the low income city of Salinas, CA; using a similar model, the investigators aim to teach research methods to a new group of Richmond youth.

ELIGIBILITY:
Inclusion Criteria:

* Household has a gas stove
* Household has a range hood that vents to the outdoors
* Household in Richmond or San Pablo

Exclusion Criteria:

* Child has other significant medical illnesses (e.g. prematurity, diabetes)
* living with a smoker who smokes indoors
* family knows they will not have stable housing for the period of the study
* Parent is not fluent in English.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Balmes, MD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share data but the investigators would be willing to entertain requests from other researchers for sharing of de-identified data only. Subjects will be asked to give permission for release of photographs of them for future presentations and other outreach materials.

REFERENCES:
- [Derived] Holm SM, Singer BC, Kang Dufour MS, Delp W, Nolan JES, Bueno de Mesquita PJ, Ward B, Williamson Y, Le O, Russell ML, Harley KG, Balmes JR. Measured air quality impacts after teaching parents about cooking ventilation with a video: a pilot study. J Expo Sci Environ Epidemiol. 2025 Apr;35(2):223-232. doi: 10.1038/s41370-024-00730-6. Epub 2024 Nov 9. PMID 39521897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment primarily occurred through East Bay pediatric clinics via recruitment fliers and information cards. At a few clinics, postcard mailings were also sent to potentially eligible patients. We also advertised for the study on an institutional website, through social media, and via fliers at community spaces (libraries, community centers, etc).
Pre-assignment Details: Due to low enrollment during the study period (height of the COVID-19 pandemic), the study shifted to a before-after trial so no group assignments were performed.
Groups:
- Intervention After 1-2 Weeks: This arm will have baseline data on air pollutant levels, stove use and range hood use collected for one week prior to receiving an educational intervention aimed at increasing use of the range hood. Data following the intervention will be collected for an additional week.
  Cooking Ventilation Intervention: An educational video presentation for the families regarding the importance of ventilation use during and after cooking, and strategies for improving the ventilation during cooking, has been created by Dr. Holm, with input from Youth Research Assistants (YRAs) The youth involvement will help to ensure that the information is presented in a way that will resonate with the local community and will also provide the youth with exposure to developing health education tools. The educational video will be shown to families at the time of the intervention visit and they will receive printed reminder materials of what they have learned.
Period: Pre-Intervention
Arm/Group | Intervention After 1-2 Weeks
Started | 19
Completed | 18
Not Completed | 1
Not completed — Intervention (hood retrofit) beyond the scope available in the study, so participation ended. | 1
Period: Post-Intervention
Arm/Group | Intervention After 1-2 Weeks
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Though 23 participants screened in for the study and consented to collection of screening data, 3 participants were unable to get initial visits scheduled in time to complete the study prior to the loss of study staff. 1 participant we stopped being able to reach. Thus, 19 were consented for the full study and began baseline.
Groups:
- Intervention After 1-2 Weeks: Baseline data on air pollutant levels, stove use and range hood use were collected for one week prior to receiving an educational intervention aimed at increasing use of the range hood. Data following the intervention will be collected for an additional 1-2 weeks.
  Cooking Ventilation Intervention: An educational video presentation for the families regarding the importance of ventilation use during and after cooking, and strategies for improving the ventilation during cooking, was been created by Dr. Holm, with input from Youth Research Assistants (YRAs). The youth involvement helped to ensure that the information was presented in a way that will resonate with the local community. The educational video was shown to families at the time of the intervention visit and they will receive printed reminder materials of what they have learned.
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8 [7.3 to 9.7]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: male | 10
  Sex: female | 13
  Sex: intersex | 0
  Sex: other | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 5
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23
Asthma Diagnosis [Count of Participants; unit: Participants]
  Ever diagnosed with asthma | 7
  Never diagnosed with asthma | 16

OUTCOME MEASURES:

1. Primary Outcome: Continuously-Measured Home PM2.5 (Fine Particulate Matter) Levels Prior to Intervention
Description: Home PM2.5 levels were measured in real-time with eLichens sensors.
Time Frame: 1-2 weeks
Measure: Median (Inter-Quartile Range); unit: (mcg/m3)*min
Groups:
- Intervention After 1-2 Weeks: This arm had baseline data on air pollutant levels, stove use and range hood use collected for one week prior to receiving an educational intervention aimed at increasing use of the range hood. Data following the intervention were collected for an additional 1-2 weeks.
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 19
(mcg/m3)*min | 10200 [275 to 65200]
Statistical Analysis 1: Comparison: Intervention After 1-2 Weeks; comparing pre and post intervention PM2.5; Test type: Other; p = 0.050, Wilcoxon Ranked Sum

2. Primary Outcome: Continuously-Measured Home PM2.5 (Fine Particulate Matter) Levels Following Intervention
Description: Home PM2.5 levels were measured in real-time using the eLichens sensors
Time Frame: 1-2 weeks
Population: 1 participant did not continue to the post-intervention interval because intervening on their home's range hood would have required resources outside the scope of the project.
Measure: Median (Inter-Quartile Range); unit: (mcg/m3)*min
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 18
(mcg/m3)*min | 4570 [0 to 31000]

3. Primary Outcome: Continuously-Measured Home NO2 (Nitrogen Dioxide) Levels Prior to Intervention
Description: Home NO2 levels were measured in real-time using eLichens sensors
Time Frame: 1-2 weeks
Measure: Median (Inter-Quartile Range); unit: ppb*min
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 19
ppb*min | 50600 [3400 to 181000]

4. Primary Outcome: Continuously-Measured Home NO2 (Nitrogen Dioxide) Level Following Intervention
Description: Home NO2 levels were measured with eLichens sensors
Time Frame: 1-2 weeks
Measure: Median (Inter-Quartile Range); unit: ppb*min
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 18
ppb*min | 15900 [3740 to 88500]
Statistical Analysis 1: Comparison: Intervention After 1-2 Weeks; comparing pre v post intervention NO2; Test type: Other; p = 0.043, Wilcoxon Ranked Sum

5. Secondary Outcome: Spirometry- Forced Vital Capacity (FVC)
Description: Spirometry is a non-invasive measure of lung function. Spirometry will be performed using an Easy One Air Spirometer; staff will be trained thoroughly in administration of the test. Forced Vital Capacity measures the total volume of air that a person can breathe out forcefully from a full breath, blowing all of it out.
  Z-Scores were created using global lung initiative normative data. A Z-score of 0 represents the population mean for a participant of that age, sex and height. A decrease in Z scores suggests worsened lung function over time.
Time Frame: measured at the end of the pre-intervention interval
Population: spirometry can be technically challenging, especially for younger children, and thus we only have results for a subset of the participants.
Measure: Median (Full Range); unit: Z-score
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 11
Z-score | 0.7 [-1.6 to 1.5]

6. Secondary Outcome: Spirometry- Forced Expiratory Volume in One Second (FEV1)
Description: Spirometry is a non-invasive measure of lung function. Spirometry will be performed using an Easy One Air Spirometer; staff will be trained thoroughly in administration of the test. Forced expiratory volume in one second measures the volume of air that a person breathes out forcefully in the first second of blowing out a full breath.
  Z-Scores were created using global lung initiative normative data. A Z-score of 0 represents the population mean for a participant of that age, sex and height. A decrease in Z scores suggests worsened lung function over time.
Time Frame: measured at the end of the pre-intervention interval
Population: these are the data for the 11 children who were able to successfully complete the spirometry maneuver, which can be conceptually challenging, especially for young children.
Measure: Median (Full Range); unit: Z-score
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 11
Z-score | 0.5 [-3.0 to 1.2]

7. Secondary Outcome: Spirometry-Forced Vital Capacity (FVC)
Description: Spirometry is a non-invasive measure of lung function. Spirometry was be performed using an Easy One Air Spirometer. Forced Vital Capacity measures the total volume of air that a person can breathe out forcefully from a full breath, blowing all of it out.
  Z-Scores were created using global lung initiative normative data. A Z-score of 0 represents the population mean for a participant of that age, sex and height. A decrease in Z scores suggests worsened lung function over time.
Time Frame: measured at the end of the post-intervention interval
Measure: Median (Full Range); unit: Z-score
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 11
Z-score | -0.3 [-1.7 to 0.8]
Statistical Analysis 1: Comparison: Intervention After 1-2 Weeks; comparing FVC pre and post intervention; Test type: Other; p = 0.056, Wilcoxon Ranked Sum

8. Secondary Outcome: Spirometry- Forced Expiratory Volume in One Second (FEV1)
Description: Spirometry is a non-invasive measure of lung function. Spirometry was performed using an Easy One Air Spirometer. Forced expiratory volume in one second measures the volume of air that a person breathes out forcefully in the first second of blowing out a full breath.
  Z-Scores were created using global lung initiative normative data. A Z-score of 0 represents the population mean for a participant of that age, sex and height. A decrease in Z scores suggests worsened lung function over time.
Time Frame: measured at the end of the post-intervention interval
Measure: Median (Full Range); unit: Z-score
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 11
Z-score | -0.5 [-2.3 to 0.7]
Statistical Analysis 1: Comparison: Intervention After 1-2 Weeks; Comparing FEV1 pre and post intervention; Test type: Other; p = 0.058, Wilcoxon Signed Rank

9. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Description: FeNO s a non-invasive measure of airways inflammation. FeNO was performed using a NIOX Vero device.
Time Frame: measured at the end of the pre-intervention interval
Population: This is again a cognitively tricky maneuver to execute, so these 9 children are those that were able to complete FeNO.
Measure: Median (Full Range); unit: ppb
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 9
ppb | 19.7 [8.0 to 53.0]

10. Secondary Outcome: Fractional Exhaled Nitric Oxide (FeNO)
Description: FeNO is a non-invasive measure of airways inflammation. FeNO will be performed using a NIOX Vero device.
Time Frame: measured at the end of the post-intervention interval
Measure: Median (Full Range); unit: ppb
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 12
ppb | 22.5 [5.0 to 60.7]
Statistical Analysis 1: Comparison: Intervention After 1-2 Weeks; comparing FeNO pre v post intervention; Test type: Other; p = 0.058, Wilcoxon Ranked Sum

11. Secondary Outcome: Asthma Control
Description: Asthma control was assessed using the widely-accepted, validated Childhood Asthma Control Test (cACT) for children with asthma.
  The cACT scale ranges from 0 to 27. Values up to 15 represent very poorly controlled asthma, 16-20 represents poorly controlled asthma and 21 or greater is considered well-controlled asthma.
Time Frame: measured at the end of the pre-intervention interval
Population: assessed only among those with asthma, and 4/4 completed the survey in this interval
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 4
score on a scale | 25 [23 to 26]

12. Secondary Outcome: Asthma Control
Description: as for outcome 11
Time Frame: measured at the end of the post-intervention interval
Population: Assessed only in those with asthma. 3/4 participants completed this survey in the post-interval.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention After 1-2 Weeks
Number analyzed (Participants) | 3
score on a scale | 26 [24 to 27]

ADVERSE EVENTS:
Time Frame: We monitored for Adverse Events from enrollment and through the over the full period of data collection which ranged from 12 to 54 days among different participants (based on changing protocols during the pandemic).
Description: No adverse events occured.
Arm/Group | Intervention After 1-2 Weeks
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04464720/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT04464720/SAP_001.pdf